CLINICAL TRIAL: NCT03475134
Title: Phase I Study to Assess Feasibility and Safety of Adoptive Transfer of Autologous Tumor-Infiltrating Lymphocytes in Combination with Interleukin-2 Followed by Nivolumab Rescue for Advanced Metastatic Melanoma
Brief Title: TIL-ACT After NMA Chemo with IL-2 and Nivo Rescue in Metastatic Melanoma (mMEL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, George Coukos, MD, PhD, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-ATATIL-2016
Record Dates: First submitted 2018-02-16; First posted 2018-03-23 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; Interleukin-2; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TIL-ACT +/- Nivolumab rescue (Experimental): Non-myeloablative lymphodepleting chemotherapy (cyclophosphamide and fludarabine), Tumor Infiltrating Lymphocyte (TIL)-Adoptive Cell Therapy (ACT), Interleukin-2 (IL-2), Nivolumab rescue
  Interventions: Other: TIL; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2; Drug: Nivolumab

INTERVENTIONS:
Other: TIL — Adoptive transfer of Autologous Tumor-Infiltrating Lymphocytes
Drug: Cyclophosphamide — Cyclophosphamide will be administered as an intravenous (IV) infusion for two days.
Drug: Fludarabine — Fludarabine will be administered as an intravenous (IV) infusion for five days.
Drug: Interleukin-2 — After TIL infusion, IL-2 (optional) will be started as a bolus administration every eight hours, for a maximum of eight doses.
Drug: Nivolumab — Nivolumab will be administered for maximum 24 months as follows: first year: 240 mg every 2 weeks; second year: 480 mg every 4 weeks.

SUMMARY:
This is a single center, single arm phase I trial to test the feasibility and safety of Tumor- Infiltrating Lymphocyte-Adoptive Cell Therapy (TIL-ACT) followed by nivolumab rescue in unresectable locally advanced or metastatic melanoma patients. The trial is based on lymphodepleting chemotherapy followed by ACT, utilizing ex vivo expanded TILs in combination with high dose interleukin-2 (IL-2) (optional, depending on patient's tolerance), followed by nivolumab rescue (if indicated) for a maximum duration of 2 years.

DETAILED DESCRIPTION:
The objective of the trial is to define the feasibility and safety of TIL-ACT in metastatic melanoma patients. In addition, the feasibility and safety of nivolumab rescue in patients with advanced metastatic disease is examined.

Study treatment will begin with intravenous non-myeloablative (NMA) lymphodepleting chemotherapy composed by fludarabine and cyclophosphamide. Both treatments will be started on the same day. Fludarabine will be administered for five days, and cyclophosphamide for two days. TILs will be infused intravenously over a period of 20-30 minutes. Between 3 and 24 hours after the infusion of TILs, optional IL-2 will be started as a bolus administration every eight hours at minimum form the start of each administration, for a maximum of eight doses, with a maximum interval of 24 hours. In order to avoid profound and long-lasting neutropenia, pegfilgrastim will be given subcutaneously. Supportive care will be given during the recovery phase from immune depletion and IL-2 therapy.

Nivolumab rescue will be initiated for eligible patients. For all patients, the first on-treatment radiological assessment will be performed 30 days after the TIL infusion, and then at month 3, and then every 12 weeks for the first 3 years of follow-up and every 4-6 months for the next 2 years, until progression.

Two Positron Emission Tomography-Computed Tomography (PET-CT) (18FDG (Fludeoxyglucose (F18)) and 68Ga-NODAGA-RGD ((68)Ga-labelled NOTA-conjugated RGD peptide) will be performed at baseline, following chemotherapy, and between 22-30 days after the TIL infusion.

The safety assessment for TIL-ACT (TLT (treatment-limiting toxicity) period) will extend from day -7 (when NMA chemo starts) till 30 days after TIL infusion.

The first three evaluable patients will be enroled no less than 2 weeks apart from each other. An interim analysis of safety at our center will be performed at the completion of the TLT period of the third evaluable patient.

ELIGIBILITY:
Inclusion criteria:

1. Patient has provided informed consent to receive TIL-ACT treatment prior to initiation of any study-specific activities/procedures.
2. Histologically confirmed diagnosis of melanoma.
3. Patients with unresectable locally advanced (stage IIIc) or metastatic (stage IV) melanoma who have progressed on at least 1 standard first line therapy, including but not limited to chemotherapy, B-Raf proto-oncogene, serine/threonine kinase (BRAF) and Mitogen-Activated Protein Kinase/Extracellular signal-Regulated Kinase (MEK) inhibitors, anti-Cytotoxic T-lymphocyte Associated 4 (CTLA4), anti-Programmed Cell Death-1 (PD-1), anti-Programmed Cell Death Ligand-1 (PD-L1) or anti-Lymphocyte-activation gene 3 (LAG3) antibodies and/or the combination.
4. Patients who have previously undergone tumor resection or biopsy and for whom pre-REP TILs are already available and adequate for further REP expansion. The following conditions have to be met:

   • The CTE GMP Manufacturing facility / sponsor representative confirms that adequate pre-REP material (in quantity and quality) is available to move to REP. In cases where more than one collected material is available for a given patient, the CTE GMP Manufacturing facility (in agreement with the sponsor) will decide which material will be used for further expansion.
5. Male or female age ≥ 18 to ≤ 70 years at the time of informed consent. Patients aged >70 will be evaluated by the investigator, and decision will be made according to patient's status, upon agreement with the PI.
6. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) of 0, 1 or 2
7. Life expectancy of greater than 12 weeks.
8. Radiologically measurable and clinically evaluable disease (as per RECIST v1.1).
9. At least one biopsiable metastatic lesion
10. In case of brain metastasis, patients must have three or fewer residual brain metastases that are less than 1 cm in diameter and asymptomatic, provided that all lesions have been adequately treated with stereotactic radiation therapy or gamma knife therapy. Lesions should be stable for 1 month, as determined by CT or MRI evaluation, after treatment and should not require steroids. Patients with surgically resected brain metastasis are eligible independently of the size of the metastasis.
11. Serology:

    * Seronegative for HIV infection (anti-HIV-1/-2)
    * Seronegative for hepatitis B infection (HBs Ag, total anti-hemoglobin C (HBc), anti-HBs). Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen HBsAg test and a positive anti-HBc antibody test) are eligible, if hepatitis B virus (HBV) DNA test is negative.
    * Seronegative for hepatitis C infection (anti-HCV): if a patient has positive anti-HCV antibody, a negative hepatitis C virus (HCV) RNA need to be obtain to register the patient.
12. Hematology

    * Absolute neutrophil count ≥ 1 x 10^9 cell/L without the support of granulocyte colony stimulating factor (G-CSF).
    * Platelet count ≥ 100 x 10^9 cell/L
    * Hemoglobin ≥ 80 g/L. Subjects may be transfused to reach this cut-off.
13. Coagulation

    * International normalization ratio (INR) or prothrombin time (PT) ≤1.5 times the upper limit of normal (x ULN) unless the subject is receiving anticoagulant therapy as long as PT and partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants.
    * PTT or activated PTT (aPTT) ≤ 1.5 x ULN unless the subject is receiving anticoagulant therapy as long as PT and PTT/aPTT is within therapeutic range of intended use of anticoagulants.
14. Chemistry:

    * Serum alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) ≤ to 3 x ULN (even in case of liver metastasis).
    * Total bilirubin ≤1.5 x ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin ≤2.5 x ULN
    * Serum creatinine ≤1.5 x ULN or creatinine clearance by Cockcroft-Gault formula ≥ 50 ml/min.
15. Adequate cardiovascular function, with documented left ventricular ejection fraction (LVEF) ≥ 45%
16. Adequate respiratory function with forced expiratory volume in 1 second (FEV1) ≥ 65% predicted, forced vital capacity (FVC) ≥ than 65% predicted and diffusing capacity of the lung for carbon monoxide (CO) (DLCO) ≥ than 50% predicted corrected.
17. At the time the patient receives the preparative regimen (NMA chemotherapy), ≥21 days must have elapsed from the time of any antibody therapy that could affect an anti-cancer immune response, including but not limited to anti-CTLA4, anti-PD-1, PD-L1 or anti-LAG3 antibody therapy or their combination.
18. Patients' toxicities from previous treatments must have recovered to a grade 1 or less according to NCI CTCAE 5.0, except for immune mediated-toxicities described below, as long as they do not put at risk the patient's condition and do not require systemic immunosuppressive steroids at immunosuppressive doses, including but not limited to:

    * Alopecia
    * Skin disorders
    * Stable neuropathy
    * Endocrinopathies requiring replacement treatment

    Note: For other medical conditions, prior discussion and agreement with the Principal Investigator is mandatory.

    Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.
19. For women of childbearing potential (WOCBP: sexually mature women who have not undergone a hysterectomy, have not been naturally post-menopausal for at least 12 consecutive months or have a serum follicle-stimulating hormone (FSH) < 40 mIU/ml (milli international units/ml)):

    * Agreement to follow instructions for contraception for the couple from screening until month number 6 of the study, in case of women not receiving nivolumab; for women receiving nivolumab, they are required to follow instructions for contraception for the couple, during participation in the trial and for the 5 months after last nivolumab infusion.
    * Negative pregnancy test (urine or serum) during screening.
20. For men participating in the trial and their female partners: agreement to follow instructions for contraception for the couple from screening until month number 6 of the study in case of patients not receiving nivolumab; when patients are receiving nivolumab, they are required to follow instructions for contraception for the couple, during participation in the trial and for the 7 months after last nivolumab infusion.

Exclusion criteria:

1. Primary uveal melanoma.
2. Patients with symptomatic and/or untreated brain metastases. Patients with definitively-treated brain metastases will be considered for enrollment after agreement with PI, as long as lesions are stable for ≥ 14 days prior to beginning the chemotherapy, there are no new brain lesions, and the patient does not require ongoing corticosteroid treatment.
3. Patients with an active second malignancy except for

   1. non-melanoma skin cancer that has been apparently cured or successfully resected
   2. carcinoma in situ as long as they have been adequately treated. Patients who have a history of malignancy are not considered to have an active malignancy if they have completed therapy and are considered by their treating investigator to be at ≤ 30% risk for relapse in 5 years following diagnosis.
4. Active systemic infections or severe infections within four weeks prior to beginning of NMA chemotherapy.
5. History of myocardial infarction or unstable angina within six months of enrolment
6. Patient requiring regular systemic immunosuppressive therapy (for example for organ transplantation, chronic rheumatologic disease); all immunosuppressive medications including but not limited to steroids, mycophenolate mofetil, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor a (TNFa) agents must have been discontinued within the last two weeks prior to starting NMA chemotherapy.

   Note: Use of inhaled or topical steroids or corticosteroid use for radiographic procedures is permitted.

   Note: The use of physiologic corticosteroid replacement therapy is permitted.
7. History of idiopathic pulmonary fibrosis or evidence of active pneumonitis (any origin)
8. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
9. History of immediate hypersensitivity reaction to aminoglycosides (e.g. gentamicin or streptomycin).
10. Participation in a research project using radiation sources exceeding an effective dose of 5mSv (milli Sievert) with no direct benefit within the 12 last months.
11. Women who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
12. Subjects for whom there are concerns that they will not reliably comply with the requirements for contraception should not be enrolled into the study.
13. Any serious underlying medical condition that could interfere with study medication.
14. Any mental or other impairment that may compromise compliance with the requirements of the study.
15. Patient participation in any other study currently receiving treatment. If the patient is in the follow-up period, he/she may be enrolled, as far as no less than 21 days have elapsed since the last previous treatment administration and the preparative regimen (NMA chemotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of TIL-ACT - successful Rapid Expansion Protocol (REP) | Evaluated for each patient at day 0 (5-10 days after chemotherapy start). After day 0 of the last patient, the number of patients with successful REP/ start of TIL-ACT infusion will be calculated.
  Number of patients for whom TIL cultures after REP achieve the required cell number and release criteria to start TIL-ACT infusion
Feasibility of TIL-ACT - successful infusion | Evaluated for each patient at day 0 (5-10 days after chemotherapy start), up to 60 mins after start of TIL-ACT infusion. At day 0 of the last patient, the number of patients with successful TIL-ACT infusion will be calculated.
  Number of patients receiving a complete TIL-ACT infusion (full NMA chemo and at least partial TIL infusion; no minimum IL-2 required)
Toxicity of TIL-ACT | 37 days after chemotherapy start (TLT period)
  Number of patients with adverse events as assessed by CTCAE version 5

SECONDARY OUTCOMES:
Feasibility of nivolumab rescue following TIL-ACT | 6 months from nivolumab start/ 100 days after end of nivolumab treatment
  Number of patients included in the 'nivolumab rescue' population
Toxicity of nivolumab rescue | 6 months from nivolumab start/ 100 days after end of nivolumab treatment
  Number of patients receiving nivolumab with adverse events as assessed by CTCAE version 5.0
Objective response rate (ORR) | 6, 12, 24, 36, 48 and 60 months
  Best overall response
Progression free survival (PFS) for TIL-ACT | 5 years
  Time from start of NMA chemotherapy until objective tumor progression (using RECIST criteria and iRECIST) or death if not documented progression.
Progression free survival (PFS) in the nivolumab rescue phase | 5 years
  Time from start of nivolumab treatment until objective tumor progression (using RECIST criteria and iRECIST) or death if not documented progression.
Overall survival (OS) | 5 years
  Time from start of NMA chemotherapy until death

OTHER OUTCOMES:
Exploratory endpoints: immune monitoring | 5 years
  Immune monitoring of the peripheral and tumor immune by Human Leukocyte Antigen (HLA) determination, immunohistochemistry, T-cell Receptor (TCR) sequencing, RNA expression and single-cell analyses, in order to correlate immune parameters in the tumor microenvironment with clinical response
Exploratory endpoints: tumor neoangiogenesis | 5 years
  Tumor neoangiogenesis using 68Ga-NODAGA-RGD PET-CT to explore correlation with clinical response
Exploratory endpoints: tumor metabolism | 5 years
  Tumor metabolism using 18FDG PET-CT to explore correlation with response to TIL-ACT

CONTACTS AND LOCATIONS:
Overall Officials: George Coukos, MD, PhD, Principal Investigator — Department director
Locations (1):
- CHUV Oncology Department, Lausanne, Canton of Vaud, Switzerland